CLINICAL TRIAL: NCT00173004
Title: Angiotensinogen Gene and Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9200200767
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2003-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Genetic studies of hypertension, focusing on renin-angiotensin system genes and other interacting genes

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension

Exclusion Criteria:

* Patients with hypertension and reluctant for the study

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ti Tsai, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan